CLINICAL TRIAL: NCT02949752
Title: Aripiprazole as an Adjunct to Atypical Antipsychotics for Weight Reduction and Improvement in Metabolic Profile
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Mental Health, Singapore (Other)
Responsible Party: Principal Investigator, Dr Bhanu Gupta, Consultant Psychiatrist, Institute of Mental Health, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 518-2015
Record Dates: First submitted 2016-10-04; First posted 2016-10-31 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Antipsychotics Weight Gain
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aripiprazole Adjunct (Experimental): Aripiprazole 5 mg as a fixed dose as adjunct to other antipsychotics
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole 5 mg every morning will be prescribed for 12 weeks

SUMMARY:
This is an open label study to prospectively evaluate the effect of adjunct use of Aripiprazole, as an agent to improve metabolic profile and induce weight loss in patients established on atypical antipsychotics (Olanzapine, Clozapine and Risperidone).

DETAILED DESCRIPTION:
The metabolic syndrome (MetS) is a well described cluster of interrelated risk factors for developing cardiovascular disease and type 2 diabetes. The main components of MetS are central obesity, hypertension, hyperglycaemia and dyslipidaemia. Individuals with MetS are two to three times more likely to have a heart attack or stroke and five times more likely to develop type 2 diabetes than those without. Metabolic abnormalities have often been identified in individuals with schizophrenia. Since the introduction of second generation antipsychotics, evidence has accumulated of their link with metabolic abnormalities. An abnormality in glucose metabolism, particularly diabetes mellitus (DM), has received the most attention. Other conditions such as cardiovascular morbidity, abnormal lipid metabolism and obesity also have a serious impact on the physical health of individuals with schizophrenia. Several pharmacological strategies are under investigation for countering the metabolic side effects, of which antipsychotic Aripiprazole has shown good evidence, when switched to as monotherapy, and also as an adjunct .

The study is planned as an open label study. An open label exploratory design will help test the hypothesis that use of adjunct Aripiprazole can help with reducing weight gain on atypical antipsychotics, and improve metabolic parameters. The number of patients in each arm is designed to yield an 80% power to detect significant differences in weight from baseline at P<0.05. There is no randomisation, blinding or placebo control, as this study is planned to test the initial hypothesis, which can inform further RCT's, if results are encouraging.

Participants will initially be screened to ensure that they fulfil the inclusion criterion, and eligible participants will be entered into the 12 week study, where they will be prescribed 5 mg Aripiprazole per day, in addition to their routine atypical antipsychotic. The typical dose range of the routine atypical antipsychotics are clozapine 200-450 mg, olanzapine 5-20mg and risperidone 2-16mg respectively. During the 12 week study, the dose of the antipsychotic and Aripiprazole should stay unchanged. If the clinical situation warrants a change in dose of antipsychotic or switch of antipsychotic, the participant will be withdrawn from the study. Atypical antipsychotic other than the ones under investigation will be prohibited, as well as medications or supplements for weight loss or weight gain, or medications known to have substantial propensity for weight changes. Benzodiazepines, anticholinergics, sleep aides will generally be allowed. Antidepressants and mood stabilisers at a stable dose, which patients were receiving prior to the study, will be allowed. Patients at high risk of suicide or self-harm as assessed by the study investigator, will be withdrawn from the study, as well as those with significant side effects from adjunct Aripiprazole.

The primary objective of the study is to assess mean change of weight from the baseline after use of adjunct Aripiprazole. The secondary endpoints include changes in metabolic parameters (waist circumference, fasting blood glucose, HbA1c, total, HDL and LDL cholesterol levels).Safety and tolerability will be measured by Simpson Angus Scale (SAS total score), Side Effects Checklist, Barnes Akathisia Scale (BAS), Abnormal Involuntary Movement Scale (AIMS), adverse events or serious adverse events reports.

The study will also evaluate neurocognition via a brief battery of 2 tests - the digit sequencing and symbol coding. These 2 tasks have been shown in a previous study to explain 76% of the variance of global neurocognition in a large sample of patients with schizophrenia. In our local sample, it was similarly shown that these 2 tasks are valid, representing 72% of the variance in global neurocognition in schizophrenia (unpublished results). The avoidance of a language component in these 2 tasks is a significant strength in choice of cognitive tasks as has been previously shown that the local population tend to underperform on language-based cognitive tasks.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patients (21 to 65 yrs)
2. Diagnosis of Schizophrenia or Schizoaffective Disorder
3. Outpatients
4. On stable doses of atypical antipsychotics, either Olanzapine, Clozapine, or Risperidone for at least 1 month
5. Patients can be on other concomitant medications. Patients can be on antipsychotic polypharmacy, but there should not be more than 1 of the above 3 atypicals in a single prescription.
6. Patients should be able to provide written informed consent.
7. Currently with a BMI ≥ 25 (Overweight) and/or ≥7% increase in weight from pre-antipsychotic treatment.

Exclusion Criteria:

1. Previous allergy to Aripiprazole/contraindication to use of Aripiprazole
2. Participants with current substance misuse, including alcohol but excluding tobacco.
3. Non-compliant with prescribed medications
4. Mental Retardation
5. Presence of any major or unstable medical or neurological illness (such as uncontrolled diabetes and hypertension).
6. Participant with an eating disorder
7. Participants with serious suicidal thoughts, or who pose a serious risk of harm to self or to others.
8. Women who are pregnant or breastfeeding
9. Severe Personality Disorder
10. Diagnosis of Hyper or Hypothyroidism; Evidence of thyroid dysfunction as evidenced by serum thyroid function tests (i.e Thyroid Stimulating Hormone and Free Thyroxine (fT4) levels > 10 % above or below the limits of the normal range
11. Use of any medication for weight loss within the past one month to the study entry
12. Clinically significant abnormalities in physical examinations, ECG or lab assessments
13. Baseline BMI < 18.5kg/m2 (cut-off point for underweight adults as per World Health Organisation guidelines)
14. Unable to read or speak English

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Mean change in body weight in kilograms | 12 weeks, assessed at baseline and at final follow up at week 12
  To assess mean change in body weight from baseline to week 12 in patients receiving adjunctive Aripiprazole to atypical antipsychotic therapy, i.e. olanzapine, clozapine, risperidone.

SECONDARY OUTCOMES:
Change in waist circumference in cm | 12 weeks, assessed at baseline and at final follow up at week 12
  To evaluate change in waist circumference from baseline to week 12
Number of participants with treatment-related adverse events as assessed by Side Effects Checklist | Checklist completed every two weeks, for the study duration of 12 weeks via Face to Face interview or Telephone contact
  To evaluate safety and tolerability data on adjunctive use of Aripiprazole using side effect checklist
Number of participants with improvement or deterioration in neuro-cognition as assessed by Digit Sequencing Test and Symbol Coding Test | 12 weeks, assessed at baseline and at final follow up at week 12
  To evaluate changes in neuro-cognition from baseline to week 12
Change in fasting plasma glucose mg/dl from baseline to week 12 | 12 weeks, assessed at baseline and at final follow up at week 12
  To evaluate change in fasting plasma glucose mg/dl from baseline to week 12
Change in Total Cholesterol, LDL and HDL Cholesterol mg/dl from baseline to week 12 | 12 weeks, assessed at baseline and at final follow up at week 12
Change in HbA1c (%) from baseline to week 12 | 12 weeks, assessed at baseline and at final follow up at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bhanu Gupta, MRCPsych, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Institute of Mental Health, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleischhacker WW, Heikkinen ME, Olie JP, Landsberg W, Dewaele P, McQuade RD, Loze JY, Hennicken D, Kerselaers W. Effects of adjunctive treatment with aripiprazole on body weight and clinical efficacy in schizophrenia patients treated with clozapine: a randomized, double-blind, placebo-controlled trial. Int J Neuropsychopharmacol. 2010 Sep;13(8):1115-25. doi: 10.1017/S1461145710000490. Epub 2010 May 12. PMID 20459883
- [Derived] Gupta B, Chee KS, Neo LQ, Tang C, Hariram J, Tan GC, Verma S, Basu S, Appan DP, Ting CC, Abdin E, Lee J. Effect of aripiprazole as an adjunct to atypical antipsychotics on weight and metabolic profile: a 12-week open-label trial. Ther Adv Psychopharmacol. 2021 Oct 9;11:20451253211046765. doi: 10.1177/20451253211046765. eCollection 2021. PMID 34646440